CLINICAL TRIAL: NCT04617652
Title: Efficacy of Magnesium Sulphate on Smoothness of Extubation in Patients Undergoing General Anaesthesia With Endotracheal Intubation: a Randomized Controlled Trial
Brief Title: Smooth Extubation With Magnesium Sulphate for General Anesthesia With Endotracheal Intubation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Atef Mohamed Sayed mahmoud, Principal investigator, Fayoum University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R142
Record Dates: First submitted 2020-10-23; First posted 2020-11-05 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Smooth Extubation
Keywords: Magnesium Sulphate; General Anesthesia; Endotracheal Intubation
MeSH Terms: interventions — Magnesium Sulfate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group M (Active Comparator): Magnesium group
  Interventions: Drug: Magnesium sulfate
- Group C (Placebo Comparator): Control group
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Magnesium sulfate — Patients will receive 1 gm of magnesium in 10 ml over 5 minutes then infusion of 1 gm in 50 ml over one hour.
  Other Names: Magnesium Group
  Arms: Group M
Drug: Normal saline — Patients will receive 10 ml of saline, then infusion of 50 ml of normal saline over one hour.
  Other Names: Placebo Group
  Arms: Group C

SUMMARY:
Tracheal extubation is a critical event in the anaesthetic management of patients undergoing general anaesthesia with endotracheal intubation for elective procedures. It the state of art to provide suitable conditions for smooth extubation and avoid coughing, bucking, straining and/or laryngospasm. Several methods have been described to provide a smooth extubation, including the use of remifentanil infusion, dexmedetomidine or fentanyl. Because of its anti-inflammatory and analgesic effects and lack of respiratory depressant actions, magnesium sulphate could be an attractive alternative.

DETAILED DESCRIPTION:
A written informed consent will be obtained from all the patients. On arrival to the preparation room intravenous cannula will be inserted, no sedation will be given. In the operating theater standard monitors, non-invasive blood pressure, oxygen saturation and electrocardiogram will be applied before induction of anesthesia, capnography after induction of anesthesia and baseline heart rate (HR), mean arterial blood pressure (MAP) and oxygen saturation (SpO2 ) will be recorded.

All patients in both groups will receive standardized anesthetic technique in the form of intravenous (i.v.) propofol 2 mg/kg, i.v. fentanyl 1-2 lg/kg and atracurium 0.5 mg/kg to facilitate endo-tracheal intubation, mechanical ventilation will be adjusted to keep end tidal carbon dioxide (EtCO2) between 30 and 35 mmHg, and all drugs will be based on ideal body weight. Isoﬂurane 1% in 50% oxygen and air, and 0.15 mg/kg atracurium every 20 min will be given for maintenance of anesthesia. Intraoperative HR, MAP, EtCO2 and SpO2 values will be recorded at 5- minute intervals till the end of operation. HR and MAP will be maintained within ±20% of the baseline values. Hypotension (deﬁned as MAP < 20% of the baseline value) will be treated by a bolus of 200 ml Ringer's solution if not responding increments of 3-9 mg ephedrine will be given. Hypertension (deﬁned as MAP > 20% of the baseline value) and/or tachycardia (deﬁned as HR > 20% of the baseline value) a supplemental dose (25-50 µg) fentanyl will be given or increasing concentration of isoﬂurane. Bradycardia (HR < 50 beat per minute) persisting for >2 min will be treated with atropine, 0.4 mg i.v. boluses. Intra-operatively i.v. ondansetron, 4 mg (Zofran, GlaxoSmithKline) will be given for prevention of postoperative nausea and vomiting. After induction of anaesthesia patients will be divided into 2 groups: group C (control group) n= 30 patients will receive 10 ml of saline, then infusion of 50 ml of normal saline over one hour. Group M (magnesium group n=30 patients) will receive 1 gm of magnesium in 10 ml over 5 minutes then infusion of 1 gm in 50 ml over one hour.

By the end of surgery isoﬂurane will be discontinued and the residual neuromuscular block will be antagonized with neostigmine 0.05 mg/kg, given with atropine 0.02 mg/kg, the endotracheal tube will be removed after return of spontaneous breathing, and the patient will obey commands in semi-sitting position, then the patient will be transferred to the post-anesthesia care unit (PACU)

ELIGIBILITY:
Inclusion Criteria:

* Elective surgeries that need endotracheal intubation.
* Duration of surgery 1-3 hours
* ASA Ⅰ-Ⅱ

Exclusion Criteria:

* Refusal of patients.
* Patients with hypersensitivity to the study drug.
* Patients with cardiac disorders, bundle branch block, hart block
* Neuromuscular disease, calcium channel blocker medication or hypermagnesemia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
smoothness of extubation | Procedure (At time of extubation)
  Smoothness of extubation Grade
  1. No coughing on endotracheal tube
  2. Coughing on the tube
  3. Vomiting
  4. Laryngospasm

SECONDARY OUTCOMES:
sedation score | 1 hrs after extubation
  Ramsey sedation score (RSS): 1 - Anxious, agitated or restless; 2 - Cooperative and oriented; 3 - Responsive to commands; 4 - Asleep, but response to light glabellar tap or loud auditory; 5 - Asleep, sluggish response to glabellar tab or auditory response; and 6 - Asleep, no response
sedation score | 1 hour after extubation
  Ramsey sedation score (RSS): 1 - Anxious, agitated or restless; 2 - Cooperative and oriented; 3 - Responsive to commands; 4 - Asleep, but response to light glabellar tap or loud auditory; 5 - Asleep, sluggish response to glabellar tab or auditory response; and 6 - Asleep, no response
heart rate | 5 minutes before induction of anathesia
  hemodynamic parameters
Mean arterial blood pressure | 5 minutes before induction of anathesia
  hemodynamic parameters
SpO2 | 5 minutes before induction of anathesia
  hemodynamic parameters
EtCO2 | 5 minutes before induction of anathesia
  hemodynamic parameters
heart rate | 5 minutes after induction of anathesia
  hemodynamic parameters
Mean arterial blood pressure | 5 minutes after induction of anathesia
  hemodynamic parameters
SpO2 | 5 minutes after induction of anathesia
  hemodynamic parameters
EtCO2 | 5 minutes after induction of anathesia
  hemodynamic parameters
heart rate | 10 minutes after induction of anathesia
  hemodynamic parameters
Mean arterial blood pressure | 10 minutes after induction of anathesia
  hemodynamic parameters
SpO2 | 10 minutes after induction of anathesia
  hemodynamic parameters
EtCO2 | 10 minutes after induction of anathesia
  hemodynamic parameters
heart rate | 15 minutes after induction of anathesia
  hemodynamic parameters
Mean arterial blood pressure | 15 minutes after induction of anathesia
  hemodynamic parameters
SpO2 | 15 minutes after induction of anathesia
  hemodynamic parameters
EtCO2 | 15 minutes after induction of anathesia
  hemodynamic parameters
heart rate | 20 minutes after induction of anathesia
  hemodynamic parameters
Mean arterial blood pressure | 20 minutes after induction of anathesia
  hemodynamic parameters
SpO2 | 20 minutes after induction of anathesia
  hemodynamic parameters
EtCO2 | 20 minutes after induction of anathesia
  hemodynamic parameters
visual analogue scale (VAS) pain score | 4 hours after extubation
  the quality of analgesia between (0-100 mm) where 0=no pain and 100 = worst comprehensible pain
visual analogue scale (VAS) pain score | 6 hours after extubation
  the quality of analgesia between (0-100 mm) where 0=no pain and 100 = worst comprehensible pain
The duration of surgery | 5 minutes after extubation
  time needed to perform surgery
Intraoperative fentanyl needed | 5 minutes after extubation
  The amount of Fentanyl given intraoperative as fentanyl will be given when either heart rate or NIBP(Non-Invasive Blood Pressure) report an increase by more than 20% of the basal records
The cumulative opioids (morphine) consumption | 6 hours after surgery
  The total amount of opioids received post operative

CONTACTS AND LOCATIONS:
Overall Officials: Atef S Khalil, MD, Principal Investigator — Fayoum University Hospitals
Locations (1):
- Fayoum University hospital, Al Fayyum, Fayoum, Madīnat Al Fayyūm, Faiyum Governorate, Egypt, Egypt